CLINICAL TRIAL: NCT03744689
Title: The Effect Of Erector Spinae Plane Block On Postoperative Pain Management In Lumbar Disc Hernia Repair Operation
Brief Title: Erector Spinae Plane Block For Lumbar Disc Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Dilek İçli, Associate professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KİA2018/440
Record Dates: First submitted 2018-11-15; First posted 2018-11-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
Keywords: Lomber disc hernia; Erector spinae plane block; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Erector Spinae Plane Block Group
  Block Drug: 0,25% bupivacaine hydrochloride (20ml) will be used for blocks
  Interventions: Procedure: Erector Spinae Plane block; Drug: Bupivacaine Hydrochloride; Device: PCA
- Control Group (Sham Comparator): Sham block will be done with serum physiologic.
  Interventions: Procedure: Sham block; Device: PCA

INTERVENTIONS:
Procedure: Erector Spinae Plane block — Erector Spinae plane block will be done according to hernia level using bupivacaine hydrochloride
  Arms: Erector Spinae Plane Block
Procedure: Sham block — Sham block will be done with serum physiologic.
  Arms: Control Group
Drug: Bupivacaine Hydrochloride — 20 ml 0,25% Bupivacaine will be used for block performances
  Arms: Erector Spinae Plane Block
Device: PCA — Intravenous morphine patient controlled analgesia device will be given to the patients postoperatively and 24 hour morphine consumption will be recorded

SUMMARY:
Pain management after lomber disc hernia repair surgery is a challenging issue for anesthetists. Erector Spinae plane block is a novel analgesic technique which could be used for this purpose. Primary aim of this double blinded randomized controlled study is to compare the analgesic efficacy of this new block technique with control group in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age 18-65 years
* Undergoing elective lomber disc hernia

Exclusion Criteria:

* obesity
* ASA III - IV
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | postoperative first 24 hour
  morphine consumptions will be recorded

SECONDARY OUTCOMES:
Numeric rating scale | postoperative first 24 hour
  Numeric rating scale for pain will be used for pain evaluation. The scale is scored in a range of 0-10 with 0 representing no pain 10 representing the highest degree of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Icli, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Derived] Yorukoglu HU, Icli D, Aksu C, Cesur S, Kus A, Gurkan Y. Erector spinae block for postoperative pain management in lumbar disc hernia repair. J Anesth. 2021 Jun;35(3):420-425. doi: 10.1007/s00540-021-02920-0. Epub 2021 Mar 22. PMID 33751203